CLINICAL TRIAL: NCT07270757
Title: Impact of Pre-Ablation Prehabilitation on Clinical Outcomes and Cardiorespiratory Fitness in Patients With Atrial Fibrillation: A Randomized Controlled Trial
Brief Title: Impact of Pre-Ablation Prehabilitation on Clinical Outcomes and Cardiorespiratory Fitness in Atrial Fibrillation Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Weizhu Ju, The First Affiliated Hospital with Nanjing Medical University, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-SR-429
Record Dates: First submitted 2025-11-26; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial Fibrillation; Cardiac rehabilitation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation Group (Experimental): Structured Prehabilitation Program for 4 weeks before ablation
  Interventions: Other: 4-week structured prehabilitation program (exercise training + psychological education)
- Usual Care Group (No Intervention): Standard Preoperative Care

INTERVENTIONS:
Other: 4-week structured prehabilitation program (exercise training + psychological education) — The prehabilitation group will receive a 4-week structured program before ablation, including:
  Individualized exercise training: Prescription based on cardiopulmonary exercise test results, including aerobic exercise (40%-60% of heart rate reserve) and resistance training
  Psychological and educational intervention: Structured education based on cognitive behavioral therapy principles, focusing on addressing kinesiophobia
  Delivery mode: Hybrid (supervised in-hospital sessions + monitored home-based sessions)
  The usual care group will receive only standard preoperative education without structured rehabilitation.
  Arms: Prehabilitation Group

SUMMARY:
The primary objective of this study is to compare the effects of a preoperative prehabilitation program versus usual care on post-procedural cardiorespiratory function and clinical outcomes in patients undergoing catheter ablation for atrial fibrillation.

DETAILED DESCRIPTION:
Background The comprehensive management of atrial fibrillation (AF) has evolved from mere rhythm control to improving patients' symptoms, functional status, and long-term prognosis. While catheter ablation effectively restores sinus rhythm, a significant clinical paradox exists: many patients fail to achieve ideal recovery in objective cardiorespiratory function and subjective quality of life even after technically successful procedures. This gap between "technical success" and "functional recovery" reveals major deficiencies in the current fragmented, procedure-centric management model.

The core of this deficiency lies in the systematic neglect of patients' physiological and psychological reserves during the perioperative period. Studies show that up to 70% of AF patients experience kinesiophobia (fear of movement), which becomes exacerbated during the perioperative period and severely hinders patients' willingness and compliance to participate in rehabilitation. Meanwhile, the high incidence of atrial arrhythmic events during the three-month post-operative "blanking period" not only increases clinical management complexity but also indirectly affects patients' functional recovery through medication adjustments and activity restrictions. These factors together form a "physiological-psychological" vicious cycle that ultimately affects patients' long-term outcomes.

Study Objectives This study aims to evaluate whether a physician-supervised structured preoperative prehabilitation program can serve as an effective integrated strategy to simultaneously improve both hard clinical outcomes and objective functional indicators in AF ablation patients.

Specific objectives include:

To evaluate the improvement effect of prehabilitation on peak oxygen uptake at 3 months post-ablation To evaluate the preventive effect of prehabilitation on atrial arrhythmic events within 90 days post-ablation To evaluate the improvement effect of prehabilitation on patient-reported outcomes (including kinesiophobia, quality of life, etc.)

Study Design This is a prospective, single-center, assessor-blinded randomized controlled trial. We plan to enroll 100 eligible patients who will be randomly allocated in a 1:1 ratio to either the prehabilitation group or the usual care group.

Interventions

The prehabilitation group will receive a 4-week structured program before ablation, including:

Individualized exercise training: Prescription based on cardiopulmonary exercise test results, including aerobic exercise (40%-60% of heart rate reserve) and resistance training Psychological and educational intervention: Structured education based on cognitive behavioral therapy principles, focusing on addressing kinesiophobia The usual care group will receive only standard preoperative education without structured rehabilitation.

Assessment and Follow-up Main assessment timepoints include baseline, 3 months post-ablation, and 6 months post-ablation.

Primary endpoints: Peak oxygen uptake, incidence of atrial arrhythmic events Secondary endpoints: Other cardiorespiratory parameters, patient-reported outcomes, clinical events Safety indicators: Adverse events, program adherence Statistical Methods Intention-to-treat analysis will be applied. Continuous variables will be analyzed using ANCOVA, categorical variables using chi-square test, and time-to-event data using Kaplan-Meier survival analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years
2. Scheduled for first AF ablation
3. NYHA class I-II
4. LVEF ≥ 50%

Exclusion Criteria:

1. Significant structural heart disease (e.g., severe valvular disease)
2. Contraindications to CPET or exercise training
3. Cognitive impairment preventing cooperation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Peak Oxygen Uptake at 3 months | 3 months post-ablation
  Measure: Cardiopulmonary exercise testing
Atrial Arrhythmic Events within 90 days | Within 90 days post-ablation
  Any atrial arrhythmic events happened within 90 days after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Please Select, China

IPD SHARING:
Plan to Share IPD: No